CLINICAL TRIAL: NCT05516420
Title: Predicting Long-term Risk of Reoperations Following Abdominal and Pelvic Surgery: a Nationwide Retrospective Cohort Study
Brief Title: Predicting Abdominal Reoperation
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: NHS Research Scotland (Other)
Responsible Party: Principal Investigator, Richard ten Broek, Principal Investigator, Radboud University Medical Center
Other Study IDs: SCARreop
Record Dates: First submitted 2022-08-17; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Surgery; Abdominal Adhesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with first abdominal surgery in Scotland between 2009 and 2011: Patients with first abdominal surgery in Scotland between 2009 and 2011

SUMMARY:
Nationwide retrospective study, to predict the risk of abdominal reoperation.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing first abdominal or pelvic surgery between June 1st 2009 and June 30th 2011 in Scotland.

Exclusion Criteria:

* Positive history for abdominal surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing first abdominal or pelvic surgery between June 1st 2009 and June 30th 2011 in Scotland.
Sampling Method: Non-Probability Sample
Enrollment: 72270 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with an abdominal reoperation in the study cohort | within 5 years postoperatively
  Number of patients undergoing a reoperation after abdominal surgery

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the Scottish National Health Service (NHS). Restrictions apply to the availability of these data, which were used under license for this study. Data derived from the analysis are available from the authors with the permission of the Scottish NHS.
  The used repository was the Safe Haven (https://shs.epcc.ed.ac.uk/2fa/scotnsh.html) from the NHS.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT05516420/Prot_SAP_000.pdf